CLINICAL TRIAL: NCT01098305
Title: Efficacy of Varenicline for Smokeless Tobacco Use in India
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Robert Schnoll, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 811047
Record Dates: First submitted 2010-03-23; First posted 2010-04-02 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-06

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine smokeless tobacco chewing tobacco varenicline
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline; Counseling; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Active Comparator)
  Interventions: Drug: Varenicline; Behavioral: Counseling
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Drug: Varenicline — Participants will be randomized to receive varenicline or placebo for 12 weeks. The dosing regimen consistent with FDA guidelines will be used: Day 1-Day 3 (0.5mg once daily); Day 4-Day 7 (0.5mg twice daily); and Day 8-Day 84 (1.0mg twice daily).
  Other Names: Chantix
  Arms: Varenicline
Behavioral: Counseling — All participants will be provided with a structured behavioral counseling program, involving 6 counseling sessions by a trained NDDTC counselor. This will be a manual-based intervention and revised as needed for cultural relevance and sensitivity by Dr. Stigler. The intervention is designed to enhance awareness of the harmful effects of smokeless tobacco, assist the person in developing skills to quit and avoid relapse, and instruct the smokeless tobacco user on medication adherence, as recommended by experts in the field.
  Other Names: Behavioral Counseling

SUMMARY:
This study, based in India, is testing the efficacy of varenicline to help smokeless tobacco users with cessation efforts.

DETAILED DESCRIPTION:
The prevalence of smokeless tobacco use in the United States is low vs. cigarette smoking, yet rates have remained constant over the past few years. In contrast, the rate of smokeless tobacco use in India is 20%. Smokeless tobacco is a carcinogenic and responsible for ~10,000 deaths/year from oral cancer in India. Unfortunately, there have been remarkably few intervention trials in India for smokeless tobacco users. To date, no trial has evaluated the new FDA approved medication, varenicline, for smokeless tobacco use. We will conduct a randomized placebo-controlled trial of varenicline for smokeless tobacco dependence at the National Drug Dependence Treatment Center (NDDTC) at the All India Institute of Medicine (AIIMS) in New Delhi with 237 smokeless tobacco users. The primary aims of this trial are to: 1) enhance research capacity at the NDDTC (i.e., train AIIMS staff to implement the behavioral counseling protocol with pharmacotherapy, data collection and management procedures); 2) assess the efficacy of varenicline for increasing biochemically confirmed 7-day point prevalence smokeless tobacco quit rates at the end-of treatment; and 3) assess longitudinal patterns of relapse and recovery following treatment with varenicline. The results of this trial may guide future investments to evaluate the efficacy of varenicline for smokeless tobacco dependence in the US, which is critical since smokeless tobacco use in the US may increase in the coming years and no approved pharmacotherapy for this drug dependence exists in the US or around the globe.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* over age 18
* used smokeless tobacco every day for the past year (confirmed with urinary cotinine)
* residing within 100km of New Dehli for the next 4 months
* interested in quitting use of smokeless tobacco.

Exclusion Criteria:

* currently enrolled or plan to enroll in another tobacco cessation program in the next 4 months
* plan to use other smoking cessation treatments in the next 4 months
* smoke cigarettes
* have current substance abuse (e.g., opioids, cocaine, marijuana) verified by urine drug screen
* have current (last 6-months) alcohol consumption that exceeds 25 standard drinks/week (if past abuse, must be symptom free for ≥ the past 12 months)
* Current use or discontinuation within last 14 days of:

  1. smoking cessation medications (bupropion, Varenicline, NRT);
  2. antipsychotics, atypicals, mood-stabilizers, anti-depressants (tricyclics, SSRIs, MAOIs), anti-panic agents, anti-obsessive agents, anti-anxiety agents, stimulants;
  3. Anti-coagulants;
  4. Daily medication for asthma or diabetes (eligible with physician approval);
* are pregnant, planning a pregnancy, or lactating
* have a history or current diagnosis of psychosis, general anxiety disorder,bipolar disorder, or schizophrenia
* have a current diagnosis of depression (if past diagnosis, must be symptom free for ≥ the past 12 months)
* have an allergy to Varenicline
* ever contemplated or attempted suicide
* have serious/unstable disease within the past 6 months (e.g., cancer [but melanoma], heart disease, HIV/AIDS)
* have a history of epilepsy or seizure disorder
* have a history or diagnosis within the last 6 months of abnormal rhythms and/or tachycardia (>100 beats/minute)
* have a history or current diagnosis of COPD; cardiovascular disease (stroke, angina); heart attack in the last 6 months; and/or uncontrolled hypertension (SBP>150 or DBP>90)16)
* have a history of kidney or liver failure
* have any medical condition or medication that could compromise safety as determined by a study physician
* cannot provide informed consent or complete the study tasks as determined by the Principal Investigator or study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- All India Institute of Medical Research, New Dehli, India

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Jhanjee S, Jain R, Jain V, Gupta T, Mittal S, Goelz P, Schnoll RA. Evaluating the Effects of Varenicline on Craving, Withdrawal, and Affect in a Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Varenicline for Smokeless Tobacco Dependence in India. J Psychoactive Drugs. 2015 Sep-Oct;47(4):325-30. doi: 10.1080/02791072.2015.1075092. Epub 2015 Aug 28. PMID 26317176

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 119 | 118
Completed | 88 | 85
Not Completed | 31 | 33
Not completed — Lost to Follow-up | 31 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 119 | 118 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (8.4) | 34.7 (9.9) | 34.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 116 | 114 | 230

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Smokeless Tobacco Abstinence Biochemically Confirmed With Urine Cotinine at the End of 12 Weeks of Treatment.
Time Frame: At the end of treatment (12 weeks)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 119 | 118
participants | 30 | 23

2. Secondary Outcome: Nicotine Withdrawal and Craving, Negative Affect, Positive Affect, and Side Effects.
Description: Side Effects
Time Frame: Ongoing throughout the treatment period (Baseline to the end of treatment, 12 weeks)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 119 | 118
participants
  sleep problems | 8 | 11
  gastrointestinal problems | 8 | 9

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/118
Other Adverse Events (participants affected / at risk) | 30/119 | 28/118
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=119) | Placebo (N=118)
abnormal dreams (Psychiatric disorders) | 7 (7) | 6 (6)
High blood pressure (Cardiac disorders) | 23 (23) | 22 (22)

LIMITATIONS AND CAVEATS:
Sample size and reduced power; lack of long-term assessments; a priori inclusion of covariates in prediction models; adherence to medication was low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes